CLINICAL TRIAL: NCT06930183
Title: Awake Thoracic Epidural Anesthesia Versus General Anesthesia in Thoracotomy: A Randomized Controlled Trial
Brief Title: Awake Thoracic Epidural Anesthesia Versus General Anesthesia in Thoracotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Elsaid Abdel Fattah, Lecturer of Anesthesia, Surgical ICU and Pain Management, Faculty of Medicine, National Cancer Institute, Cairo University, Egypt., Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP2411-501-086-193
Record Dates: First submitted 2025-03-28; First posted 2025-04-16 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Awake; Thoracic Epidural Anesthesia; General Anesthesia; Thoracotomy
MeSH Terms: interventions — Bupivacaine; Anesthesia, General; Fentanyl

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Awake thoracic epidural anesthesia group (Experimental): Patients will preoperatively receive awake thoracic epidural anesthesia.
  Interventions: Drug: Awake thoracic epidural anesthesia
- General anesthesia group (Active Comparator): Patients will receive general anesthesia.
  Interventions: Drug: General anesthesia

INTERVENTIONS:
Drug: Awake thoracic epidural anesthesia — Patients will preoperatively receive awake thoracic epidural anesthesia.
  Other Names: Bupivacaine
  Arms: Awake thoracic epidural anesthesia group
Drug: General anesthesia — Patients will receive general anesthesia.
  Other Names: Fentanyl
  Arms: General anesthesia group

SUMMARY:
This study aims to compare awake thoracic epidural anesthesia and general anesthesia in thoracotomy.

DETAILED DESCRIPTION:
The severity of acute postoperative pain is a causative factor for chronic postsurgical pain, and it has been observed that the incidence of chronic postsurgical pain is very high after thoracotomy. Effective management of acute post-operative pain is a must in these patients.

Thoracic epidural analgesia (TEA) is used as an adjunct to general anesthesia (GA) in thoracic surgery. However, tthe horacic epidural blockade has been rarely utilized as a sole method to provide anesthesia for major thoracic procedures

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 75 years old.
* Both genders.
* American Society of Anesthesiologists (ASA) physical status classification II or III.
* Scheduled for thoracotomy.

Exclusion Criteria:

* Difficult airway management,
* Hemodynamically unstable patients, obesity (body mass index >30).
* Absolute contraindication to thoracic epidural anesthesia such as (patient refusal, allergy to local anesthetics, coagulopathy, active neurologic disorders, skin infection at insertion site, uncooperative patients, uncontrolled cough, and unfavorable anatomy for thoracic epidural).
* Neurological disorders: risk of seizure, unable to cooperate, intracranial mass or brain edema, extensive pleural adhesions or previous pulmonary resections, hypoxemia (PaO2 <60) or hypercarbia (PaCO2 >50)
* Poor cardiac function (ejection fraction less than 50%).
* Patients with bad pulmonary function tests.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Assessment the change in pulmonary function | 24 hours postoperatively
  The change in pulmonary function will be assessed using Forced vital capacity (FVC) will be recorded.

SECONDARY OUTCOMES:
Heart rate | Till the end of surgery (Up to 2 hours)
  Heart rate will be recorded at baseline, and every 15min till the end of surgery.
Mean arterial pressure | Till the end of surgery (Up to 2 hours)
  Mean arterial pressure will be recorded at baseline, and every 15min till the end of surgery.
Degree of pain | 48 hours postoperatively
  The patients will be instructed how to report pain by means of the visual analogue scale (VAS), in which 0 = "no pain" and 10 = "worst possible pain". VAS will be assessed at post-anesthesia care unit (PACU), 1, 2, 4, 8, 12,18, 24, 36, 48 hours postoperative.
Total morphine consumption | 48 hours postoperatively
  Rescue analgesia of morphine will be given as 3 mg bolus if the VAS > 3 to be repeated after 30 min if pain persists until the visual analogue scale (VAS) < 4.
Time to 1st rescue analgesia | 48 hours postoperatively
  Time to 1st rescue analgesia (time from end of surgery to first dose of morphine administrated).
Incidence of adverse events | 48 hours postoperatively
  Incidence of adverse events such as nausea, vomiting, and respiratory depression will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.